CLINICAL TRIAL: NCT05193214
Title: An Open Label, Single-arm Phase II Clinical Study Evaluating the Efficacy and Safety of Recombinant Anti-PD-1 Humanized Monoclonal Antibody Injection (609A) in Patients With Unresectable or Advanced Undifferentiated Pleomorphic Sarcoma
Brief Title: A Phase II Study for 609A in the Treatment of Advanced Undifferentiated Pleomorphic Sarcoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-609-UPS-II-01
Record Dates: First submitted 2021-12-31; First posted 2022-01-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: Sarcoma, Soft Tissue
Keywords: Sarcoma, Soft Tissue; 609A
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 609A UPS (Experimental): The 609A single-drug regimen (200mg Q3W) was used to treat unresectable or advanced undifferentiated pleomorphic sarcoma to evaluate the safety and effectiveness of 609A.
  Interventions: Drug: Recombinant anti-PD-1 humanized monoclonal antibody injection

INTERVENTIONS:
Drug: Recombinant anti-PD-1 humanized monoclonal antibody injection — Each subject received 609A 200 mg intravenous infusion, once every 3 weeks (Q3W), until disease progression, intolerable toxicity, death, informed withdrawal, early withdrawal from the study, loss to follow-up, or the end of the study, whichever occurs first Whichever prevails.
  Other Names: 609A

SUMMARY:
The main purpose of this study is to evaluate the efficacy and safety of recombinant anti-PD-1 humanized monoclonal antibody injection (609A) in patients with unresectable or advanced undifferentiated pleomorphic sarcoma

DETAILED DESCRIPTION:
This is a multi-center, open label, phase II clinical study. The safety and effectiveness of 609A in the treatment of unresectable or advanced undifferentiated pleomorphic sarcoma are mainly evaluated by ORR (based on the results of CT/MRI examination of subjects during treatment).

ELIGIBILITY:
Inclusion Criteria:

* A Chinese citizen who understands and is willing to sign an informed consent form (ICF).
* Age ≥18 years old and ≤75 years old, regardless of gender.
* For patients with unresectable or advanced undifferentiated pleomorphic sarcoma confirmed by cytology or histopathology, the subject is willing to provide a sufficient number of tumor tissue sections for pathological type confirmation in the central pathology room.
* At least one anthracycline-containing chemotherapy regimen failed (disease progression or intolerable toxicity).
* There is at least one measurable lesion (see RECIST 1.1 standard for definition).
* The Eastern Cooperative Oncology Group (ECOG) score 0-1 points.
* Life expectancy ≥ 3 months.
* The pregnancy test of female patients with fertility is negative within 3 days before the first administration; any male and female patients with fertility must agree to use medical approval during the entire trial period and within 6 months after the last trial drug is administered. Method of contraception.
* Before 609A starts treatment, it must have sufficient organ functions, including: a) Bone marrow reserve: absolute neutrophil (ANC) ≥1.0×10^9/L; platelet count ≥90×10^9/L; Hemoglobin ≥90g/L or ≥5.6mmol/L; b) Total bilirubin≤1.5×ULN, AST and/or ALT≤3×ULN (if abnormal liver function is caused by tumor liver metastasis, then AST and/or ALT≤5×ULN); c) Serum creatinine ≤1.5×ULN or estimated creatinine clearance ≥50mL/min (Cockroft and Gault formula); d) Coagulation test international normalized ratio (INR) ≤2 (except: warfarin anticoagulation The treated patients can receive INR 2 to ≤3), and activated partial thromboplastin time (APTT) ≤1.5×ULN.

Exclusion Criteria:

* Known to be allergic to protein drugs or recombinant proteins or excipients in 609A pharmaceutical preparations, or have severe allergic reactions after administration of other monoclonal antibodies, or have a history of life-threatening allergies.
* Have received any of the following anti-tumor treatments in the past: a) Have received any anti-tumor treatment within 4 weeks before the first administration, including chemotherapy, radiotherapy, targeted therapy, immunotherapy, hormone therapy (hormone replacement therapy, testosterone or (Except for oral contraceptives), biological therapy and anti-tumor Chinese medicine treatment, etc.; b) Have received immunoagonist treatment within 4 weeks before the first administration; c) Have previously received immunotherapy for T cell co-stimulation or checkpoint approach.
* According to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0, any residual AE from previous anti-tumor therapy did not return to grade 0 or 1, or did not meet other selections/exclusions other than this one The level specified in the standard, except for residual hair loss effects.
* Have received other drug clinical trial treatment or interventional device clinical trial treatment within 4 weeks before the first administration.
* Underwent major surgery within 21 days before the first administration.
* Live attenuated vaccine was vaccinated within 28 days before the first dose.
* Use of leukocyte-promoting factors such as granulocyte colony stimulating factor (G-CSF) or granulocyte-macrophage colony stimulating factor (GM-CSF) within 72 hours before the first administration, or 2 weeks before the first administration Have used erythropoietin (EPO) or suspended red blood cell transfusion, or have taken corrective measures such as platelet transfusion within 1 week before the first administration.
* Subjects with central nervous system (CNS) metastasis.
* Suffer from other active malignant tumors within 5 years or at the same time. Excludes cured localized tumors, such as skin basal cell carcinoma, skin squamous cell carcinoma, superficial bladder cancer, prostate carcinoma in situ, cervical carcinoma in situ, breast carcinoma in situ, etc.
* A history of any type of primary immunodeficiency, a history of stem cell or organ transplantation.
* Subjects with a history of active autoimmune diseases or autoimmune diseases, including but not limited to immune-related neurological diseases, multiple sclerosis, autoimmune (demyelinating) neuropathy, Green- Barre syndrome, myasthenia gravis, systemic lupus erythematosus (SLE), connective tissue disease, scleroderma, inflammatory bowel disease including Crohn's disease and ulcerative colitis, hepatitis, toxic epidermal necrolysis ( TEN), Stevens-Johnson syndrome (SJS) or antiphospholipid syndrome.
* Patients who need to be treated with glucocorticoid (>15mg/d prednisone or equivalent dose of hormone) or other immunosuppressive agents within 14 days before the first administration of the planned trial drug. In the absence of active autoimmune diseases, inhaled or topical glucocorticoids can be used. Hormone replacement therapy doses ≤ 10 mg/d prednisone equivalent are acceptable. Accepts ophthalmology, nasal cavity and intra-articular injection of glucocorticoids.
* There are clinically important cardiovascular and cerebrovascular diseases, including: a) Severe or uncontrollable heart disease that requires treatment, congestive heart failure The New York Heart Association (NYHA) is classified as III or IV, and drugs cannot be controlled. Stable angina pectoris, history of myocardial infarction in the past 6 months, QTc interval of electrocardiogram: male ≥450 milliseconds, female ≥470 milliseconds, severe arrhythmia requiring medical treatment (except for atrial fibrillation or paroxysmal supraventricular tachycardia) . b) Patients with indwelling heart stent within 6 months. c) Insufficient control of hypertension, systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg.
* People with a history of interstitial lung disease, idiopathic pulmonary fibrosis, unresolved active or chronic inflammatory lung disease cannot be included in the group. Subjects who have radiation pneumonia but have recovered can be included in the group;
* People with any of the following infections: a) Active hepatitis B or C. Hepatitis B virus (HBV) carriers without active disease or cured hepatitis C can be included in the group; b) Human immunodeficiency virus (HIV) infection; c) Severe chronic or active infection, requiring systemic antibacterial, antifungal or antibacterial Viral therapy, including active tuberculosis infection, etc.; d) Febrile neutropenia or unexplained single fever> 38.5°C within 1 week before the first administration of the test drug The fever generated by the tumor can be included in the group).
* Any other serious illnesses (for example: uncontrolled diabetes, active gastric ulcer, uncontrolled epilepsy, cerebrovascular events, gastrointestinal bleeding, coagulopathy with severe symptoms and signs), mental, psychological, Family or geographic conditions, based on the judgment of the investigator, may interfere with trial planning, treatment, and follow-up, or affect the subject's compliance, or put the subject at high risk of treatment-related complications.
* Women who are pregnant or breastfeeding.
* Any other situation where the investigator judges that the patient is not suitable for entry into this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-25 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR,Objective response rate | up to 18 months.
  CT/MRI examinations were performed every 6 weeks, and the efficacy of anti-tumor treatment was evaluated by RECEIST and iRECEIST standards.

SECONDARY OUTCOMES:
AE | up to 18 months.
  All adverse events related to 609A observed through various tests (including blood routine, pregnancy test, electrocardiogram, etc.)
BOR, Best overall response | up to 18 months.
  CT/MRI examinations were performed every 6 weeks, and the efficacy of anti-tumor treatment was evaluated by RECEIST and iRECEIST standards.
DCR, Disease control rate | up to 18 months.
  CT/MRI examinations were performed every 6 weeks, and the efficacy of anti-tumor treatment was evaluated by RECEIST and iRECEIST standards.
DOR, Duration of Response | up to 18 months.
  CT/MRI examinations were performed every 6 weeks, and the efficacy of anti-tumor treatment was evaluated by RECEIST and iRECEIST standards.
TTR, Time to response | up to 18 months.
  CT/MRI examinations were performed every 6 weeks, and the efficacy of anti-tumor treatment was evaluated by RECEIST and iRECEIST standards.
SD duration | up to 18 months.
  CT/MRI examinations were performed every 6 weeks, and the efficacy of anti-tumor treatment was evaluated by RECEIST and iRECEIST standards.
Immunogenicity of 609A | up to 18 months.
  Detect the presence of anti-609A antibodies through the subject's blood sample

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohui Niu, Master, Principal Investigator — Beijing Jishuitan Hospital
Locations (1):
- Beijing Jishuitan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No